CLINICAL TRIAL: NCT01247350
Title: A Single- and Multiple-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY3009104 in Japanese Healthy Subjects
Brief Title: A Study of LY3009104(Baricitinib) for Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14089; I4V-JE-JADM (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-11-17; First posted 2010-11-24 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2017-09

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 2 mg LY3009104 (Cohort 1) (Experimental): 2mg administered once on day 1 (single dose)
  Interventions: Drug: LY3009104
- 5 mg LY3009104 (Cohort 2) (Experimental): 5mg administered once on day 1 (single dose)
  Interventions: Drug: LY3009104
- 10 mg LY3009104 (Cohort 3) (Experimental): 10 mg administered on day 1 (single dose) and following a 7 day washout period, administered once daily for 10 days (multiple dose)
  Interventions: Drug: LY3009104
- 14 mg LY3009104 (Cohort 4 ) (Experimental): 14 mg administered on day 1 (single dose) and following a 7 day washout period, administered once daily for 10 days (multiple dose)
  Interventions: Drug: LY3009104
- Placebo (Placebo Comparator): administered on day 1 (single dose) and following a 7 day washout period, administered once daily for 10 days (multiple dose)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3009104 — Administered orally
  Other Names: baricitinib
  Arms: 10 mg LY3009104 (Cohort 3); 14 mg LY3009104 (Cohort 4 ); 2 mg LY3009104 (Cohort 1); 5 mg LY3009104 (Cohort 2)
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of LY3009104 when given orally as single and multiple doses in Japanese healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females. Male subjects: Agree to use 2 forms of highly effective methods of birth control with female partners of childbearing potential for the specified duration. Female subjects: Females must not be pregnant, breastfeeding, or at risk to become pregnant during study participation. Female subjects of childbearing potential must test negative for pregnancy at screening and agree to use 2 forms of highly effective methods of birth control, or remain abstinent for the specified duration.
* Up to third generation Japanese, that is defined as all of the subject's biological grandparents are of exclusive Japanese decent and have been born in Japan.
* Are between the body mass index (BMI) of 18.0 and 30.0 kg/m², inclusive at screening.

Exclusion Criteria:

* Are subjects who have previously completed or withdrawn from this study or any other study investigating LY3009104, and received the study drug.
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Show evidence of significant active neuropsychiatric disease.
* Have current or recent history of herpes zoster or simplex in the last 90 days prior to randomization, or history of herpes zoster, such as disseminated herpes zoster involving multiple dermatomes, ocular involvement, including herpes zoster involving the ophthalmic branch of the trigeminal nerve.
* Have or have a history of rheumatoid arthritis.
* History of malignancy, with the exception of cured basal cell or squamous cell carcinoma of the skin.
* History of stomach or intestinal surgery, except that appendectomy and/or cholecystectomy will be allowed.
* Receipt of blood products within 2 months prior to study entry.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 2 mg LY3009104 (Baricitinib): 2 mg administered orally once on Day 1 (single dose)
- 5 mg LY3009104: 5 mg administered orally once on Day 1 (single dose)
- 10 mg LY3009104: 10 mg administered orally on Day 1 (single dose) and following a 7-day washout period, administered once daily for 10 days ((multiple dose)
- 14 mg LY3009104: 14 mg administered orally on Day 1 (single dose) and following a 7-day washout period, administered once daily for 10 days (multiple dose)
- Placebo: administered orally on Day 1 (single dose) and following a 7-day washout period, administered once daily for 10 days (multiple dose)
Period: Overall Study
Arm/Group | 2 mg LY3009104 (Baricitinib) | 5 mg LY3009104 | 10 mg LY3009104 | 14 mg LY3009104 | Placebo
Started | 6 | 6 | 6 | 7 | 9
Received Multiple Doses of Study Drug | 0 | 0 | 6 | 6 | 5
Completed | 6 | 6 | 5 | 6 | 8
Not Completed | 0 | 0 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Not completed — Entry criteria not met | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 2 mg LY3009104: 2 mg administered orally once on Day 1 (single dose)
- Total: Total of all reporting groups
Arm/Group | 2 mg LY3009104 | 5 mg LY3009104 | 10 mg LY3009104 | 14 mg LY3009104 | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 9 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (10.8) | 48.0 (15.0) | 46.7 (9.0) | 51.1 (6.3) | 45.1 (10.7) | 47.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 2 | 2 | 12
  Male | 3 | 4 | 3 | 5 | 7 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 6 | 6 | 7 | 9 | 34
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 6 | 7 | 9 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Effects
Description: Adverse events were considered clinically significant effects. A summary of serious adverse events and other nonserious adverse events are located in the Reported Adverse Event section.
Time Frame: Days 1-10 for Cohorts 1 & 2, Days 1-7 for single dose of Cohorts 3 & 4, Days 8-31 for multiple doses
Population: Participants who were administered study drug.
Measure: Count of Participants; unit: Participants
Groups:
- 2 mg LY3009104 Single Dose: 2 mg administered orally once on Day 1
- 5 mg LY3009104 Single Dose: 5 mg administered orally once on Day 1
- 10 mg LY3009104 Single Dose: 10 mg administered orally once on Day 1
- 14 mg LY3009104 Single Dose: 14 mg administered orally once on Day 1
- Placebo Single Dose: administered orally once on Day 1
- 10 mg LY3009104 Multiple Dose: Following a 7-day washout period, participants in the 10 mg LY3009104 single-dose group received 10 mg LY3009104 once daily for 10 days
- 14 mg LY3009104 Multiple Dose: Following a 7-day washout period, participants in the 14 mg LY3009104 single-dose group received 14 mg LY3009104 once daily for 10 days
- Placebo Multiple Dose: Following a 7-day washout period, participants in the placebo single-dose group received placebo once daily for 10 days.
Arm/Group | 2 mg LY3009104 Single Dose | 5 mg LY3009104 Single Dose | 10 mg LY3009104 Single Dose | 14 mg LY3009104 Single Dose | Placebo Single Dose | 10 mg LY3009104 Multiple Dose | 14 mg LY3009104 Multiple Dose | Placebo Multiple Dose
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 9 | 6 | 6 | 5
Participants
  Serious Adverse Events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nonserious Adverse Events | 1 | 1 | 2 | 7 | 6 | 5 | 4 | 2

2. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY3009104
Description: Cmax of Day 1 is Cmax after single dose, and Cmax of Day 17 is Cmax at steady-state.
Time Frame: Day 1 and Day 17: predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
Population: Participants who were administered study drug and had pharmacokinetics (PK) samples for the analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles/Liter (nmol/L)
Groups:
- 2 mg LY3009104 Day 1: 2 mg administered orally once on Day 1
- 5 mg LY3009104 Day 1: 5 mg administered orally once on Day 1
- 10 mg LY3009104 Day 1: 10 mg administered orally once on Day 1
- 14 mg LY3009104 Day 1: 14 mg administered orally once on Day 1
- 10 mg LY3009104 Day 17: Following a 7-day washout period, participants in the 10 mg LY3009104 single-dose group received 10 mg LY3009104 once daily for 10 days
- 14 mg LY3009104 Day 17: Following a 7-day washout period, participants in the 14 mg LY3009104 single-dose group received 14 mg LY3009104 once daily for 10 days
Arm/Group | 2 mg LY3009104 Day 1 | 5 mg LY3009104 Day 1 | 10 mg LY3009104 Day 1 | 14 mg LY3009104 Day 1 | 10 mg LY3009104 Day 17 | 14 mg LY3009104 Day 17
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 5 | 6
nanomoles/Liter (nmol/L) | 76.1 (29) | 220 (35) | 327 (43) | 410 (19) | 319 (30) | 439 (9)

3. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve (AUC) of LY3009104
Description: AUC is the measure of total plasma exposure of a drug over a given time period. AUC of Day 1 is AUC from 0 to 24 hours. AUC of Day 17 is AUC during one dosing interval at steady-state.
Time Frame: Day 1 and Day 17: predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
Population: Participants who were administered study drug and had pharmacokinetics (PK) samples for the analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles*hour/Liter (nmol*h/L)
Arm/Group | 2 mg LY3009104 Day 1 | 5 mg LY3009104 Day 1 | 10 mg LY3009104 Day 1 | 14 mg LY3009104 Day 1 | 10 mg LY3009104 Day 17 | 14 mg LY3009104 Day 17
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 5 | 6
nanomoles*hour/Liter (nmol*h/L) | 403 (10) | 1240 (23) | 1730 (21) | 2790 (14) | 1970 (18) | 3060 (17)

4. Secondary Outcome: Pharmacokinetics: Half-Life(t1/2) of LY3009104
Description: Half life (t1/2) is the time measured for the plasma concentration of LY3009104 to decrease by one half.
Time Frame: Day 1 and Day 17: predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
Population: Participants who were administered study drug and had pharmacokinetics (PK) samples for the analyses.
Measure: Geometric Mean (Full Range); unit: hour (h)
Arm/Group | 2 mg LY3009104 Day 1 | 5 mg LY3009104 Day 1 | 10 mg LY3009104 Day 1 | 14 mg LY3009104 Day 1 | 10 mg LY3009104 Day 17 | 14 mg LY3009104 Day 17
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 5 | 6
hour (h) | 5.19 [3.88 to 6.31] | 6.82 [5.70 to 7.79] | 6.43 [4.37 to 9.90] | 8.48 [6.95 to 10.8] | 8.57 [7.43 to 9.30] | 9.41 [7.24 to 13.1]

5. Secondary Outcome: Pharmacokinetics: Apparent Volume of Distribution of LY3009104
Description: Apparent volume of distribution is used to quantify the distribution of a drug between plasma and the rest of the body after dosing. It is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Day 1, it is apparent volume of distribution during the terminal phase after single dose. Day 17, it is apparent volume of distribution during the terminal phase at steady-state.
Time Frame: Day 1 and Day 17: predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
Population: Participants who were administered study drug and had pharmacokinetics (PK) samples for the analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | 2 mg LY3009104 Day 1 | 5 mg LY3009104 Day 1 | 10 mg LY3009104 Day 1 | 14 mg LY3009104 Day 1 | 10 mg LY3009104 Day 17 | 14 mg LY3009104 Day 17
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 5 | 6
Liter (L) | 96.3 (18) | 99.4 (29) | 138 (41) | 150 (19) | 169 (24) | 167 (23)

6. Secondary Outcome: Pharmacokinetics: Apparent Total Body Clearance of LY3009104
Description: Apparent total body clearance is the volume of plasma from which the drug is completely removed in a given time period. For Day 1, it is apparent total body clearance of drug after single dose. For Day 17, it is apparent total body clearance of drug at steady-state.
Time Frame: Day 1 and Day 17: predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 38 and 48 hours postdose
Population: Participants who were administered study drug and had pharmacokinetics (PK) samples for the analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/h)
Arm/Group | 2 mg LY3009104 Day 1 | 5 mg LY3009104 Day 1 | 10 mg LY3009104 Day 1 | 14 mg LY3009104 Day 1 | 10 mg LY3009104 Day 17 | 14 mg LY3009104 Day 17
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 5 | 6
Liter/hour (L/h) | 12.9 (11) | 10.1 (22) | 14.8 (20) | 12.2 (17) | 13.7 (18) | 12.3 (17)

7. Secondary Outcome: Pharmacokinetics: Time of Maximum Observed LY3009104 Concentration (Tmax)
Description: Tmax is time to reach maximum observed drug concentration. For Day 1, it is tmax after single dose. For Day 17, it is tmax at steady-state.
Time Frame: Day 1 and Day 17: predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 38 and 48 hours postdose
Population: Participants who were administered study drug and had pharmacokinetics (PK) samples for the analyses.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | 2 mg LY3009104 Day 1 | 5 mg LY3009104 Day 1 | 10 mg LY3009104 Day 1 | 14 mg LY3009104 Day 1 | 10 mg LY3009104 Day 17 | 14 mg LY3009104 Day 17
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 5 | 6
hour (h) | 1.00 [0.50 to 2.00] | 1.00 [0.50 to 1.00] | 1.25 [0.50 to 2.00] | 1.00 [0.50 to 2.10] | 1.00 [0.50 to 2.00] | 1.00 [1.00 to 1.00]

8. Secondary Outcome: Pharmacokinetics: Renal Excretion of LY3009104
Description: Percentage of LY3009104 excreted in urine from zero to 24 hours.
Time Frame: Day 1: continuous for 24 hours
Population: Participants who were administered study drug (10 mg and 14 mg LY3009104 per protocol) and had pharmacokinetics (PK) samples for the analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of drug
Groups:
- 10 mg LY3009104 Day 1: 10 mg administered orally on Day 1
- 14 mg LY3009104 Day 1: 14 mg administered orally on Day 1
Arm/Group | 10 mg LY3009104 Day 1 | 14 mg LY3009104 Day 1
Number analyzed (Participants) | 6 | 7
percentage of drug | 75.8 (7) | 63.6 (13)

ADVERSE EVENTS:
Time Frame: From starting of the dose to follow-up. Adverse events (AE) for single dose were observed from Day 1 to Day 10±2 days (Cohorts 1&2) or Day 7 (Cohorts 3&4). AE for multiple doses were observed from Day 8 to Day 31±3 days.
Groups:
- 2 mg LY3009104 - Single Dose: 2 mg administered orally once on Day 1
- 5 mg LY3009104 - Single Dose: 5 mg administered orally once on Day 1
- 10 mg LY3009104 - Single Dose: 10 mg administered orally on Day 1
- 14 mg LY3009104 - Single Dose: 14 mg administered orally on Day 1
- Placebo - Single Dose: administered orally on Day 1
- 10 mg LY3009104 - Multiple Dose: Following a 7-day washout period, participants in the 10 mg LY3009104 single-dose group received 10 mg LY3009104 once daily for 10 days
- 14 mg LY3009104 - Multiple Dose: Following a 7-day washout period, participants in the 14 mg LY3009104 single-dose group received 14 mg LY3009104 once daily for 10 days
- Placebo - Multiple Dose: Following a 7-day washout period, participants in the placebo single-dose group received placebo once daily for 10 days.
Arm/Group | 2 mg LY3009104 - Single Dose | 5 mg LY3009104 - Single Dose | 10 mg LY3009104 - Single Dose | 14 mg LY3009104 - Single Dose | Placebo - Single Dose | 10 mg LY3009104 - Multiple Dose | 14 mg LY3009104 - Multiple Dose | Placebo - Multiple Dose
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/7 | 0/9 | 0/6 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 2/6 | 7/7 | 6/9 | 5/6 | 4/6 | 2/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mg LY3009104 - Single Dose (N=6) | 5 mg LY3009104 - Single Dose (N=6) | 10 mg LY3009104 - Single Dose (N=6) | 14 mg LY3009104 - Single Dose (N=7) | Placebo - Single Dose (N=9) | 10 mg LY3009104 - Multiple Dose (N=6) | 14 mg LY3009104 - Multiple Dose (N=6) | Placebo - Multiple Dose (N=5)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application Site Reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vessel Puncture Site Haematoma (General disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oral Herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Reticulocyte Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dizziness Postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days